CLINICAL TRIAL: NCT01216436
Title: Phase 1 Study of Local Modulation of Immune Receptor Function to Enhance Immune Responses to Dendritic Cell Vaccination in Subjects With Metastatic Melanoma
Brief Title: Local Modulation of Immune Receptors to Enhance the Response to Dendritic Cell Vaccination in Metastatic Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The PI retired
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None
Other Study IDs: Pro00019239
Record Dates: First submitted 2010-02-01; First posted 2010-10-07 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2014-04

CONDITIONS: Metastatic Melanoma
Keywords: melanoma; immunotherapy; dendritic cell; GITR-ligand; CTLA-4
MeSH Terms: conditions — Melanoma; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Vaccination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vaccine plus untransfected DC (Experimental): Subjects in all study arms will be vaccinated with mature autologous dendritic cells transfected with a combination of RNAs encoding melanoma tumor associated antigens MART, Tyrosinase, gp100, and MAGE-3. In this Study Arm (Study Arm A), each subject will be coinjected with additional mature autologous dendritic cells that are not transfected with RNA.
  Interventions: Biological: Vaccination with RNA-transfected mature autologous DC
- Vaccine plus GITRL RNA DC (Experimental): Subjects in all study arms will be vaccinated with mature autologous dendritic cells transfected with a combination of RNAs encoding melanoma tumor associated antigens MART, Tyrosinase, gp100, and MAGE-3. In this Study Arm (Study Arm B), each subject will be coinjected with additional mature autologous dendritic cells transfected with RNA encoding the immune modulator GITR-L.
  Interventions: Biological: Vaccination with RNA-transfected mature autologous DC
- Vaccine plus antiCTLA4 RNA DC (Experimental): Subjects in all study arms will be vaccinated with mature autologous dendritic cells transfected with a combination of RNAs encoding melanoma tumor associated antigens MART, Tyrosinase, gp100, and MAGE-3. In this Study Arm (Study Arm C), each subject will be coinjected with additional mature autologous dendritic cells transfected with RNA encoding immune modulator anti-CTLA4 mAb.
  Interventions: Biological: Vaccination with RNA-transfected mature autologous DC
- Vaccine plus GITRL/ antiCTLA4 RNA DC (Experimental): Subjects in all study arms will be vaccinated with mature autologous dendritic cells transfected with a combination of RNAs encoding melanoma tumor associated antigens MART, Tyrosinase, gp100, and MAGE-3. In this Study Arm (Study Arm D), each subject will be coinjected with additional mature autologous dendritic cells transfected with RNA encoding both GITR-L and anti-CTLA4 mAb immune modulators.
  Interventions: Biological: Vaccination with RNA-transfected mature autologous DC

INTERVENTIONS:
Biological: Vaccination with RNA-transfected mature autologous DC — Dendritic cells (DC) will be administered at a dose of 20 million cells by intranodal injection under ultrasound guidance. Each subject will receive a total of six vaccinations at one week intervals

SUMMARY:
Our proposed study is designed to test the safety of a new vaccine against melanoma. The induction of immune activity against cancers such as melanoma is a promising approach to cancer treatment, but to date, only a few clinically significant immune responses have been seen following vaccine therapy. This is an important problem, since there are very limited treatment options for patients with metastatic melanoma (melanoma that has spread to lymph nodes and organs).

Studies suggest that monoclonal antibodies (mAbs) that block inhibitory receptors on immune cells can enhance the immune responses against cancer, but the intravenous injection of such mAbs has caused severe side effects in animals and humans. In our laboratory, we have developed a method to deliver mAbs and other proteins that block such inhibitory receptors locally at the site where immune responses against melanoma proteins are stimulated by vaccination, enhancing anti-melanoma immunity while avoiding the side-effects associated with intravenous injection of these immune modulators. This is achieved by loading dendritic cells, a type of immune cell, with RNA that encodes the immune modulator. The RNA-loaded dendritic cells then make the immune modulatory proteins and release them locally. By mixing these dendritic cells with additional dendritic cells loaded with melanoma proteins, the immune modulators are released at the site where anti-melanoma immune cells are stimulated.

In this phase I trial, subjects with metastatic melanoma will undergo the process of leukapheresis, in which white blood cells are removed from the body. Monocytes, a type of immune cell, will then be purified from the white blood cells and cultured under conditions that will change them into dendritic cells. Half of these dendritic cells are then loaded with melanoma antigen RNA, which will lead to the production of melanoma antigen proteins within the dendritic cells. The remaining half of the dendritic cells will be either untreated or loaded with RNA encoding immune modulators so that these dendritic cells will release immune modulators at the site of vaccination. These dendritic cells will be mixed with the melanoma antigen-loaded dendritic cells and injected as a vaccine into lymph nodes. Each subject will receive six weekly injections of their own dendritic cells. Safety and toxicity will be closely monitored. In addition, immune responses against melanoma, as well as clinical responses, will be assessed.

DETAILED DESCRIPTION:
A variety of trials of immunotherapy in metastatic melanoma have clearly demonstrated that immune responses against melanoma can be induced, but only a few patient have responded clinically, suggesting that new strategies to enhance anti-cancer immune responses are needed. Most of these immunotherapy trials have focused on antigen delivery and providing stimulatory antigen-specific signals to T cells. However, the induction of antigen-specific T cell-mediated immune responses is regulated not only by stimulatory signals, but also by inhibitory receptor-mediated signals. Studies have demonstrated that administering mAbs targeting such immune-modulating receptors on T cells enhances vaccine-induced anti-tumor immunity, suggesting that such an approach might improve the efficacy of clinical cancer vaccines. However, systemic administration such mAbs has been associated with severe, sometimes fatal, autoimmunity. We have developed an approach for targeted delivery of such immune modulatory proteins and mAbs, using immune modulator RNA-transfected dendritic cells (DC), to sites where anti-tumor T cells are induced. Our preliminary studies indicate that this approach may eliminate the adverse effects associated with systemic administration immune modulators, while also enhancing vaccine-induced immune responses.

Therefore, the objective of this proposed Phase I immunotherapy trial is to determine the safety and obtain preliminary data on the efficacy of vaccination of human subjects with melanoma tumor associated antigen (TAA) RNA-transfected mature monocyte-derived DC coadministered with additional untransfected DC (Study Arm A), DC transfected with RNA encoding a soluble GITR-L fusion protein (Study Arm B), DC transfected with RNA encoding the humanized heavy and light chains of an antagonistic anti-CTLA-4 mAb (Study Arm C), or DC transfected with combined GITR-L and anti-CTLA-4 mAb RNA (Study Arm D). All study subjects will undergo leukapheresis for collection of peripheral blood mononuclear cells (PBMC) and purified monocytes will be cultured with the cytokines GM-CSF and IL-4 to produce immature DC. After the induction maturation with a standard cytokine cocktail, half of the DC will then be transfected with RNA encoding melanoma TAAs MART, tyrosinase, and gp100, and MAGE-3, while the remaining half of the DC will be either untransfected (Study Arm A) or will be transfected with immune modulator RNA (Study Arm B, C, and D). DC will be cryopreserved. Subjects will then be immunized with these DC, weekly for six intranodal injections. For each subject, safety and toxicity will be assessed, and anti-tumor immune responses will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed metastatic melanoma
* Karnofsky performance status greater than or equal to 70%.
* Estimated life expectancy > 6 months.
* Age > 17 years.
* Adequate hematologic function with:

  * WBC >= 3000 mm3
  * hemoglobin >= 9 mg/dl
  * platelets >= 100,000/mm3
* Adequate renal and hepatic function with:

  * serum creatinine < 2.5 mg/dl
  * bilirubin < 2.0 mg/dl
  * AST/SGOT < 70 U/L
  * ALT/SGPT < 70 U/L
  * Alkaline Phosphatase ≤ 135 U/L
* Ability to understand and provide signed informed consent that fulfills Institutional Review Board guidelines.
* Ability to return to Duke University Medical Center for adequate follow-up as required by this protocol.

Exclusion Criteria:

* Subjects undergoing concurrent chemotherapy, radiation therapy, or immunotherapy will be excluded.
* The subject has previously irradiated, surgically treated, or newly diagnosed central nervous system (CNS) metastases will be excluded (Pre-enrollment head CT is not required if not indicated by clinical signs or symptoms).
* Subjects with a history of autoimmune disease such as, but not restricted to, inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis will be excluded.
* Subjects with serious concurrent chronic or acute illness such as pulmonary (asthma or COPD), cardiac (NYHA class III or IV) or hepatic disease, or other illness considered by the principal investigator to constitute an unwarranted high risk for investigational drug administration will be excluded.
* Subjects with medical or psychological impediment to probable compliance with the protocol will be excluded.
* Subjects with concurrent second malignancy other than melanoma or non-melanoma skin cancer will be excluded. In the event of prior non-melanoma malignancies treated surgically, the subject must be considered NED (no evidence of disease) for a minimum of 3 years prior to enrollment.
* Presence of an active acute or chronic infection, including symptomatic urinary tract infection, HIV (as determined by ELISA and confirmed by Western Blot) or viral hepatitis (as determined by HBsAg and Hepatitis C serology) will lead to subject exclusion.
* Subjects receiving steroid therapy (or other immunosuppressive agents such as azathioprine or cyclosporine A) are excluded on the basis of potential immune suppression.
* Subjects with inadequate peripheral vein access to undergo leukapheresis will be excluded.
* Female subjects with a positive pregnancy test, as well as those who have not previously undergone hysterectomy and/or bilateral oophorectomy and are unwilling to utilize a medically approved form of contraception, from the time of enrollment until 6 weeks after the final immunization, will be excluded.
* Male subjects, not previously surgically sterilized, who are unwilling to use a condom with spermicide during any sexual activity occurring over the entire immunization period and for the 6 weeks that immediately follow the final immunization will be excluded.
* Subjects with a documented history of severe allergic reaction to beta-lactams, eggs or soy products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | A minimum of 6 months
  Safety and Tolerability will be assessed for all subjects during the vaccination period and then regularly during the post-vaccination period. All subjects will then be followed clinically as would be done any subject with melanoma for a total of 5 years.

SECONDARY OUTCOMES:
Cellular anti-melanoma immune responses will be assessed | A minimum of 4 months
  T cells from blood collected after each vaccination and following the full course of vaccination will be assessed for melanoma antigen-specificity using Interferon-gamma Elispot and cytotoxicity assays. Immune responses will be assessed following each vaccination and then will continue to be assessed until anti-melanoma immune responses return to baseline levels.

CONTACTS AND LOCATIONS:
Overall Officials: Scott K Pruitt, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Pruitt SK, Boczkowski D, de Rosa N, Haley NR, Morse MA, Tyler DS, Dannull J, Nair S. Enhancement of anti-tumor immunity through local modulation of CTLA-4 and GITR by dendritic cells. Eur J Immunol. 2011 Dec;41(12):3553-63. doi: 10.1002/eji.201141383. Epub 2011 Oct 26. PMID 22028176
- [Background] Boczkowski D, Lee J, Pruitt S, Nair S. Dendritic cells engineered to secrete anti-GITR antibodies are effective adjuvants to dendritic cell-based immunotherapy. Cancer Gene Ther. 2009 Dec;16(12):900-11. doi: 10.1038/cgt.2009.39. Epub 2009 Jun 5. PMID 19498460